CLINICAL TRIAL: NCT01075659
Title: Nicotine Pharmacodynamics With a New Oral Nicotine Replacement Product and NiQuitin™ Lozenge: A Study in Healthy Smokers
Brief Title: Early Effects of a New Oral Nicotine Replacement Product and NiQuitin™ Lozenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NICTDP2011
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation; VAS; Urges to smoke
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LHN1548 (Experimental): Two single doses of an experimental Nicotine Replacement Therapy (NRT) 2 mg, with five hours between treatments. Seven hours duration of total follow-up period.
  Interventions: Drug: Nicotine
- 2019706 (Active Comparator): Two single doses of Nicotine Lozenge 2 mg, with five hours between treatments. Seven hours duration of total follow-up period.
  Interventions: Drug: Nicotine
- 2020005 (Active Comparator): Two single doses of Nicotine Lozenge 4 mg, with five hours between treatments. Seven hours duration of total follow-up period.
  Interventions: Drug: Nicotine

INTERVENTIONS:
Drug: Nicotine — Two single doses of experimental Nicotine Replacement Therapy (NRT) 2 mg, with five hours between treatments. Seven hours duration of total follow-up period
  Other Names: Not yet marketed
  Arms: LHN1548
Drug: Nicotine — Two single doses of Nicotine Lozenge 2 mg, with five hours between treatments. Seven hours duration of total follow-up period.
  Other Names: NiQuitin™ lozenge 2 mg
  Arms: 2019706
Drug: Nicotine — Two single doses of Nicotine Lozenge 4 mg, with five hours between treatments. Seven hours duration of total follow-up period.
  Other Names: NiQuitinTM lozenge 4 mg
  Arms: 2020005

SUMMARY:
A comparison of two products for oral nicotine replacement with respect to relief of urges to smoke after single doses of nicotine.

DETAILED DESCRIPTION:
This study compares a new oral Nicotine Replacement Therapy (NRT) product with NiQuitin™ lozenge 2 mg and 4 mg, respectively, after 5 hours of witnessed nicotine abstinence with respect to urges to smoke during the first 5 minutes after start of treatment. Single doses of each treatment are given during separate treatment visits scheduled in a crossover setting with randomized treatment sequences. The study will include 200 healthy smokers between 19-55 years, who have been smoking at least 10 cigarettes daily during at least one year preceding inclusion, and who smoke within 30 minutes of waking up. Subjects, study personnel and monitor will be aware of what type of product is administered at a given visit, but not of the administered dose of the lozenge.

ELIGIBILITY:
Inclusion Criteria:

* Healthy smokers, smoking at least 10 cigarettes daily during at least one year preceding inclusion, and smoking within 30 minutes of waking up.
* Female participants of child-bearing potential are required to use a medically acceptable means of birth control.
* A personally signed and dated informed consent document, indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Pregnancy, lactation or intended pregnancy.
* Use of NRT, bupropion, or varenicline, or history of a quit attempt later than 3 months before screening visit.
* Treatment with an investigational product, other than those described in the protocol, between 1 month preceding the first treatment visit and the last treatment visit of the study.
* Prior regular use of any of the investigational products.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Areas under the linearly interpolated urges to smoke vs. time curve evaluated in a hierarchical order starting with the 5 minutes' evaluation (AUC5min, AUC3min, AUC1min) | from time zero following 5 hours of smoking abstinence (baseline), until 5 minutes, until 3 minutes, and until 1 minute, respectively

SECONDARY OUTCOMES:
Areas under the linearly interpolated urges to smoke vs. time curve (AUC10min) | from time zero following 5 hours of smoking abstinence (baseline), until 10 minutes thereafter
Time to a 25%, 50%, 75%, and 90% reduction from baseline intensity of urges to smoke score | from time zero following 5 hours of smoking abstinence (baseline), until 2 hours thereafter
Proportion of subjects reaching 25%, 50%, 75% and 90% reduction of urges to smoke | from time zero following 5 hours of smoking abstinence (baseline), until 2 hours thereafter
Study treatment acceptability, evaluated using pair-wise treatment comparisons of ordered categorical-scale assessments | At the end of three separate visits, at least 36 hours apart

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- Clinical Pharmacology, Lund, Sweden